CLINICAL TRIAL: NCT01091363
Title: A Randomized Controlled Clinical Trial of a Combination of Pharmacotherapy and Culturally Tailored Cognitive Behavior Therapy With Korean Americans
Brief Title: Tobacco Dependence Treatment for Asian Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Sun S Kim, Study Principle Investigator, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5K23DA021243-02 (NIH)
Record Dates: First submitted 2010-03-21; First posted 2010-03-24 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Tobacco Dependence
Keywords: smoking cessation; tobacco dependence treatment; cultural adaptation; Asian Americans
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- deep cultural arm (Experimental): deep cultural therapy
  Interventions: Behavioral: Deep Cultural
- standard arm (Active Comparator): brief cessation counseling
  Interventions: Behavioral: Standard

INTERVENTIONS:
Behavioral: Standard — 10 minute brief cessation counseling
  Arms: standard arm
Behavioral: Deep Cultural — Deep culturally tailored cognitive behavioral therapy
  Arms: deep cultural arm

SUMMARY:
Nicotine dependence is very common among Asian Americans; yet, research on understanding and treating nicotine dependence in this group is almost nonexistent. The proposed study is a first attempt to develop a smoking cessation program that is tailored to Korean-culture specific aspects. It is proposed that Korean Americans who receive a culturally tailored smoking cessation program will be more likely to have prolonged abstinence at 12-month follow-up than their counterparts who receive brief cessation counseling. Subjects in both arms receive nicotine patches for 8 weeks. Self-reported abstinence is validated with exhaled carbon monoxide and salivary cotinine tests.

DETAILED DESCRIPTION:
Korean men have been known for very high smoking rates and the highest cancer death smoking-attributable fraction. In contrast, Korean women reportedly smoke at low rates compared to the general U.S. population. However, recent population-based survey data indicate steady increases in smoking prevalence of Korean American women. Particularly, it has been found that they tend to initiate smoking as they acculturate into social norms of American women. Preliminary data of the applicant and others suggests interventions must be culturally adapted and a motivation-based and family-involved approach is most promising. The training plan will help the applicant develop an independent program of drug abuse research that focuses on better understanding and treating tobacco dependence among Asian Americans, including evaluating culturally competent and gender-specific interventions. The research plan will examine the impact of culture and gender on nicotine dependence and utilize National Institute on Drug Abuse behavioral therapy development methods. The proposed research plan has two-phases and evaluates tobacco dependence treatment with Korean Americans (N = 164, 50% women). Phase 1 is a no-control group study (Stage Ia) that is aimed at developing an intervention manual of Group-based Motivational Interviewing (GMI) intervention, therapists' adherence and competence scales, training program, and small feasibility intervention study with 20 Korean-American (offered separately for men and women). Phase 2 is a randomized controlled trial (Stage Ib) with 144 Korean Americans that is conducted to assess feasibility and relative effectiveness of the GMI behavioral intervention in conjunction with Nicotine Replacement Therapy (NRT) in comparison with a brief group medication management of NRT. Gender-interaction effects of psychosocial variables on treatment outcomes will be assessed, including acculturation and depression. This award will help prepare the applicant for an independent research career focusing on Asian Americans and Nicotine Dependence, including adapting and testing new interventions for different populations.

ELIGIBILITY:
Inclusion Criteria:

Korean-speaking Koreans who:

1. Are ages of 18 and older
2. Have been smoking at least 10 or more cigarettes on average per day for the past 30 days; AND
3. Are willing to quit smoking and receive NRT

Exclusion Criteria:

1. Inability to speak and understand Korean or English
2. Involvement in behavioral or other pharmacological smoking cessation programs
3. History of serious cardiac diseases and/or presence of skin diseases (see Human Subjects); OR
4. Pregnancy, lactation or plans to become pregnant in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun S Kim, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, the data will be sent.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: October 2009-September 2016
Access Criteria: Researchers at non-profit academic institutions
URL: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4250475/pdf/nihms-600738.pdf

REFERENCES:
- [Result] Kim SS, Kim SH, Ziedonis D. Tobacco dependence treatment for Korean Americans: preliminary findings. J Immigr Minor Health. 2012 Jun;14(3):395-404. doi: 10.1007/s10903-011-9507-0. PMID 21785963
- [Result] Kim SS, Kim SH, Fang H, Kwon S, Shelley D, Ziedonis D. A Culturally Adapted Smoking Cessation Intervention for Korean Americans: A Mediating Effect of Perceived Family Norm Toward Quitting. J Immigr Minor Health. 2015 Aug;17(4):1120-9. doi: 10.1007/s10903-014-0045-4. PMID 24878686
- [Derived] Kim SS, Fang H, Bernstein K, Zhang Z, DiFranza J, Ziedonis D, Allison J. Acculturation, Depression, and Smoking Cessation: a trajectory pattern recognition approach. Tob Induc Dis. 2017 Jul 24;15:33. doi: 10.1186/s12971-017-0135-x. eCollection 2017. PMID 28747857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2010-2013.
Pre-assignment Details: 232 people were screened and 123 were excluded before randomization.
Groups:
- Deep Cultural: This arm received eight weekly 40-minute individualized counseling sessions of cognitive behavioral therapy and cultural tailoring intervention (CBCT) plus 8-week NRT
  nicotine patch: 8-week nicotine patch therapy
- Standard: This arm received eight, weekly 10-minute brief cessation counseling sessions that are not tailored to Korean culture.
  nicotine patch: 8-week nicotine patch therapy
Period: Overall Study
Arm/Group | Deep Cultural | Standard
Started | 55 | 54
Completed | 42 | 37
Not Completed | 13 | 17
Not completed — Withdrawal by Subject | 11 | 15
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Smokers of Korean ethnicity residing in the United States
Groups:
- Deep Cultural: eight weekly 40-minute individualized counseling sessions of cognitive behavioral therapy and cultural tailoring intervention (CBCT) plus 8-week NRT
  nicotine patch: 8-week nicotine patch therapy
- Standard: This arm receives eight, weekly 10-minute brief cessation counseling sessions that are not tailored to Korean culture.
  nicotine patch: 8-week nicotine patch therapy
- Total: Total of all reporting groups
Arm/Group | Deep Cultural | Standard | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 105
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — age at the time of study enrollment
  years | 50.69 (8.41) | 48.76 (10.08) | 49.73 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 46 | 45 | 91
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: 12-month Abstinence
Description: The number of participants who had maintained smoking abstinence for the past 12 months
Time Frame: 12 months
Population: Korean Americans
Measure: Count of Participants; unit: Participants
Groups:
- Cultural Tailoring; Brief Cessation Counseling: The 12-month prolonged abstinence was defined as being continuously abstinent from the quit day except for the first 2-week grace period. Self-reported abstinence was biochemically verified with expired-air CO (< 6 parts ppm) and saliva cotinine (≤ 30ng/ml) tests. We used a Micro+ Smokerlyzer CO Monitor (Bedfont Scientific, NJ) and NicAlert® test strips.
Arm/Group | Cultural Tailoring | Brief Cessation Counseling
Number analyzed (Participants) | 55 | 54
Participants | 21 | 6
Statistical Analysis 1: Comparison: Cultural Tailoring vs Brief Cessation Counseling; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 4.67, 95% CI 2-sided [1.67 to 12.99]

2. Secondary Outcome: Perceived Family Norm Toward Quitting Smoking
Description: Perceived family norm toward quitting smoking was assessed using the Perceived Family Norm Index consisting of two items assessing normative beliefs (i.e., "I believe that my family [my friends] wants me to quit smoking") and motivation to comply with the belief (i.e., "I am willing to comply with the belief"). Score for each item can range from -3 "strongly disagree" to +3 "strongly agree". The total score is the sum of the scores of the two items and can range from -6 to +6.
Time Frame: 6-month follow-up
Population: Korean Americans
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cultural Tailoring | Brief Cessation Counseling
Number analyzed (Participants) | 55 | 54
score on a scale | 5.14 [3 to 6] | 4.81 [2 to 6]
Statistical Analysis 1: Comparison: Cultural Tailoring vs Brief Cessation Counseling; Mediation analyses were performed to examine the effect of the intervention on abstinence via the three theoretic variables (attitudes, perceived family norms, and self-efficacy), using the Hayes' PROCESS computation tool for a serial multiple mediator model with a binary outcome variable (quitting vs. smoking); Test type: Superiority or Other — Hayes' PROCESS computation tool for a serial multiple mediator model predicting a binary logistic outcome; p = 0.02, Mediation Analysis; Mean Difference (Net) = 1.92, 95% CI 2-sided [0.34 to 6.32]

3. Other Pre Specified Outcome: Biochemical Verification of Self-reported Abstinence
Description: The salivary cotinine level was assessed by a NicAlert® test, using adopted a cutoff level 2 (30-100ng/ml).
Time Frame: 12-month follow-ups
Population: Korean Americans who had smoked at least 10 cigarettes a day for the past 6 months before study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cultural Tailoring | Brief Cessation Counseling
Number analyzed (Participants) | 55 | 54
Participants | 21 | 6

ADVERSE EVENTS:
Time Frame: 1 year
Description: There was no case of participants at risk for other adverse events.
Groups:
- Cultural Tailoring: The group who received a deep Korean-culture tailored smoking cessation intervention.
- Brief Cessation Counseling: The group who received a standard non-culture tailored smoking cessation intervention.
Arm/Group | Cultural Tailoring | Brief Cessation Counseling
Serious Adverse Events (participants affected / at risk) | 3/55 | 2/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cultural Tailoring (N=55) | Brief Cessation Counseling (N=54)
skin reaction (Skin and subcutaneous tissue disorders) | 3/3 (3) | 2/2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No